CLINICAL TRIAL: NCT05181514
Title: Impact of Plasma Lipids on β Cell Function and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Full Professor, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Intralipid01
Record Dates: First submitted 2021-12-06; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Hypertriglyceridemia; Glucose Intolerance
MeSH Terms: conditions — Hypertriglyceridemia; Glucose Intolerance | interventions — soybean oil, phospholipid emulsion; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Placebo Comparator): Participants will undergo a dual labeled, 3-h oral glucose tolerance test (OGTT) during i.v. infusion of normal saline
  Interventions: Other: Normal Saline
- 20% Intralipid (Experimental): Participants will undergo a dual labeled, 3-h oral glucose tolerance test (OGTT) during i.v. infusion of Intralipid 20%.
  Interventions: Other: 20% Intralipid

INTERVENTIONS:
Other: 20% Intralipid — Participants will receive a 5 h primed (375 mL/m2)-continuous (25 mL h-1 m-2) i.v. infusion of 20% fat emulsion (Intralipid 20%), together with a 5 h primed (28 µmol/kg)-continuous (0.28 µmol min-1 kg-1) infusion of 6,6-[2H2]glucose. After 2 h, participants will consume within 5 min an oral glucose drink consisting of 147 mL of 50% dextrose solution (wt/vol) enriched with 1.5 g of [U-13C] glucose.
  Arms: 20% Intralipid
Other: Normal Saline — Participants will receive a 5 h primed (375 mL/m2)-continuous (25 mL h-1 m-2) i.v. infusion of normal saline (Sodium Chloride 0.9%), together with a 5 h primed (28 µmol/kg)-continuous (0.28 µmol min-1 kg-1) infusion of 6,6-[2H2]glucose. After 2 h, participants will consume within 5 min an oral glucose drink consisting of 147 mL of 50% dextrose solution (wt/vol) enriched with 1.5 g of [U-13C] glucose.
  Arms: Normal Saline

SUMMARY:
The investigators aim to evaluate whether and to what extent glucose tolerance, beta cell function, insulin clearance, and glucose metabolic fluxes change in response to an acute increase in plasma triglycerides during lipid infusion, independently of free fatty acid (FFA) levels, in nondiabetic subjects.

DETAILED DESCRIPTION:
Mild hypertriglyceridemia is associated with reduced glucose tolerance and increased risk of type 2 diabetes, independent of obesity, in both cross-sectional and prospective studies. It is unclear whether this association is direct or mediated by circulating lipid substrates of triglycerides (free fatty acids, or FFA) and which are the mechanisms involved.

To comprehensively examine the effects of mild acute hypertriglyceridemia on major glucose homeostatic mechanisms involved in diabetes progression, two dual-labeled oral glucose tolerance tests (OGTT) during 5-hour intravenous infusions of either 20% Intralipid or normal saline will be performed in healthy lean volunteers. Lipid-induced changes in glucose tolerance and insulin metabolism will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* Body mass index (BMI) 18-35 kg/m2
* both women and men

Exclusion Criteria:

* chronic or acute diseases
* any medications
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Glucose control | At the end of the 5-hour lipid infusion
  Incremental area under the curve (AUC) of plasma glucose in response to the oral glucose tolerance test (OGTT)
Insulin secretion | At the end of the 5-hour lipid infusion
  Insulin secretion rate (ISR) estimated from C-peptide deconvolution at fasting and in response to the oral glucose tolerance test (OGTT)
Beta cell glucose sensitivity | At the end of the 5-hour lipid infusion
  Beta cell glucose sensitivity calculated by mathematical modeling of insulin secretion rate (ISR) and plasma glucose concentrations during the oral glucose tolerance test (OGTT)
Insulin sensitivity | At the end of the 5-hour lipid infusion
  Insulin sensitivity estimated by an OGTT-derived surrogate index (Matsuda index)
Insulin clearance | At the end of the 5-hour lipid infusion
  Insulin clearance calculated as the ratio between insulin secretion rate (ISR) and plasma insulin levels
Rate of oral glucose appearance (RaO) | At the end of the 5-hour lipid infusion
  The rate of oral glucose appearance (RaO) will be assessed from the time course of the plasma tracer/tracee ratio of 6,6-[2H2]glucose and [U-13C]glucose
Endogenous glucose production (EGP) | At the end of the 5-hour lipid infusion
  The endogenous glucose production (EGP) will be assessed from the time course of the plasma tracer/tracee ratio of 6,6-[2H2]glucose and [U-13C]glucose

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, MD, Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No